CLINICAL TRIAL: NCT02576327
Title: A Multi-central Perspective Randomized Controlled Study Evaluating the Efficacy and Safety of Aprepitant in Autologous Hematopoietic Stem Cell Transplantation
Brief Title: A Study Evaluating the Efficacy and Safety of Aprepitant in Autologous Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jun Zhu (Other)
Responsible Party: Sponsor-Investigator, Jun Zhu, Department of Hematology Oncology, clinical oncology college, Director of department, Party Secretary, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-2015YJZ25
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Vomiting
Keywords: Lymphoma; Aprepitant; Chemotherapy-induced nausea and vomiting (CINV); Autologous Hematopoietic Stem Cell Transplantation; Hematological Malignancies
MeSH Terms: conditions — Vomiting; Lymphoma; Hematologic Neoplasms | interventions — Tropisetron; Dexamethasone; dexamethasone 21-phosphate; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant Arm (Experimental): Tropisetron 5mg（Day1-6）+ Dexamethasone 10mg（Day1-6）+ Aprepitant125mg（Day1-2）、80mg（Day3-6）
  Interventions: Drug: Tropisetron; Drug: Dexamethasone; Drug: Aprepitant
- Control Arm (Active Comparator): Tropisetron 5mg（Day1-6）+ Dexamethasone 10mg（Day1-6）
  Interventions: Drug: Tropisetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Tropisetron — Tropisetron Hydrochloride Injection 5mg (Day 1-6)
  Other Names: Tropisetron Hydrochloride Injection
Drug: Dexamethasone — Dexamethasone Sodium Phosphate Injection 10mg (Day 1-6)
  Other Names: Dexamethasone Sodium Phosphate Injection
Drug: Aprepitant — Aprepitant 125mg （Day1-2）, 80mg (Day 3-6)
  Other Names: Emend
  Arms: Aprepitant Arm

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of additional aprepitant to standard antiemetic regimen in Autologous Hematopoietic Stem Cell Transplantation.

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) is a serious complication of treatments of hematological malignancies. Although aprepitant has been shown to control CINV in highly emetogenic therapies for solid tumors, the antiemetic effect of aprepitant in hematological chemotherapies is still not clear. In this multi-central perspective randomized controlled study, the investigators are trying to evaluate the efficacy and safety of additional aprepitant to standard antiemetic regimen in Autologous Hematopoietic Stem Cell Transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >/= 18 years, <65 years
* Patients with lymphoma receiving autologous hematopoietic stem cell transplantation for the first time
* ECOG 0-2
* TBIL,AST and ALT < 2.5-fold upper normal range
* Female and male subjects of childbearing potential must agree to use a medically accepted method of adequate contraception.
* Signed informed consent

Exclusion Criteria:

* Prior autologous/ allogeneic hematopoietic stem cell transplantation for lymphoma
* Women who are pregnant or breast feeding.
* Serious or uncontroled infection
* Serious complications
* Severe renal or hepatic disease
* Severe mental or nervous system diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall complete response (no emesis and no rescue therapy) | During and post chemotherapy (0-120 h)

SECONDARY OUTCOMES:
Time to initial neutrophil engraftment | 30 days post-transplantation
  Time to initial neutrophil engraftment is defined as 1st of 3 consecutive days of an ANC ≥0.5 × 10^9/L
Time to initial platelet recovery | 30 days post-transplantation
  Time to initial platelet recovery is defined as 1st of 3 consecutive platelet count measurements tested on different days with a count ≥20 × 10^9/L with no platelet transfusion in the prior 7 days.
Quality of Life | During and post chemotherapy (0-120 h)
Safety and Tolerability assessed by possible side effects, and all AE will be reported during 30 days after the chemotherapy. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute